CLINICAL TRIAL: NCT06981065
Title: The Scandinavian Displaced Lateral Clavicle Trial (ScanDiLaC) - A Multicentre, Pragmatic, 12-Month, Non-inferiority, Randomized Controlled Trial
Brief Title: The Scandinavian Displaced Lateral Clavicle Trial
Acronym: ScanDiLaC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01097-01
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Clavicle Fracture
Keywords: Displaced lateral clavicle fracture; Non-surgical; Surgical; PROMs; Health economy; Non-inferior; Complications
MeSH Terms: interventions — Physical Therapy Modalities; Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Parallell with cross-over option in non-surgical arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-surgical (Experimental): Non-surgical treatment with a simple sling and physiotherapy. Cross-over option at 6 weeks if signs of symptomatic delayed union, non-decreasing pain, and patient requests surgery
  Interventions: Procedure: Simple Sling and Physiotherapy
- Surgical (Active Comparator): Surgical treatment with plate and screws
  Interventions: Procedure: Surgical treatment

INTERVENTIONS:
Procedure: Simple Sling and Physiotherapy — Non-surgical treatment with a simple sling and physiotherapy according to standardized program.
  Arms: Non-surgical
Procedure: Surgical treatment — Surgical treatment with plate and screws (lateral clavicle plate, clavicle plate or hook plate with/without coracoclavicular fixation).
  Arms: Surgical

SUMMARY:
A multicentre multinational RCT to investigate whether non-surgical treatment is non-inferior to surgical treatment for displaced extraarticular lateral clavicle fractures in adults.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether non-surgical treatment is non inferior to surgical treatment for displaced lateral clavicle fractures with regards to functional outcome measured with different patient-reported outcome measures. Patients aged 18-65 years will be randomized to non-surgical or surgical (pragmatic) treatment. The primary outcome is the Disabilities of Arm Hand and Shoulder (DASH) score at 1 year.

ELIGIBILITY:
Inclusion Criteria:

- Displaced extraarticular lateral clavicle fracture (type II or V according to the modified Neer classification)

Exclusion Criteria:

* Pathological fracture
* Open fracture
* Neurovascular injury
* Same-time fracture in the upper extremity
* Polytrauma
* Contraindications to surgery and/or anesthesia
* Unable to give informed consent
* Inability to complete follow-up

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Disabilites of the Arm, Shoulder and Hand (DASH) | 1 year
  A 30-item patient-reported outcome measure concerning shoulder, arm and hand function, with two additional 4-item modules concerning work and sports function.
  Min: 0 Max: 100. 0 representing no disability and 100 representing the most severe disability. A DASH score of 50 or more is often considered a cutoff for the presence of severe disability, while 20 or more suggests a medium level of disability.

SECONDARY OUTCOMES:
Disabilites of the Arm, Shoulder and Hand (DASH) | Pre-injury, 6 weeks, 3 months, 6 months, 2 years, 5 years
  A 30-item patient-reported outcome measure concerning shoulder, arm and hand function, with two additional 4-item modules concerning work and sports function.
  Min: 0 Max: 100 0 representing no disability and 100 representing the most severe disability. A DASH score of 50 or more is often considered a cutoff for the presence of severe disability, while 20 or more suggests a medium level of disability.
Nottingham Clavicle Score (NCS) | 6 weeks, 3 months, 6 months, 1, 2, 5 years
  A 10-item disease-specific PROM concerning functional outcome after injuries and diseases around the clavicle.
  The minimum possible score is 20, and the maximum is 100. A higher score indicates better functional ability, while a lower score suggests greater functional disability. The NCS can be graded as excellent (80-100), good (60-79), fair (40-59), or poor (<40).
University of California, Los Angeles (UCLA) Activity scale | Pre-injury, 6 weeks, 3 months, 6 months, 1 years
  An activity scale measured in 10 levels. It ranges from 1 to 10, with 1 representing no physical activity and 10 representing regular participation in impact sports.
EuroQol 5-Dimension 5-Level (EQ-5D-5L) questionnaire | Pre-injury, 6 weeks, 3 months, 6 months, 1, 2, 5 years
  Health-Related Quality of Life (HRQoL) measured in 5 Levels. The minimum and maximum possible outcomes for EQ-5D-5L index scores are -0.573 and 1, respectively. The minimum value represents a health state considered worse than death, while 1 represents full health.
Visual Analog Scale (VAS) for pain | Baseline, 6 weeks, 3 months, 6 months, 1, 2, 5 years
  Pain measure by visual analog scale in 11 levels. Minimum 0 and maximum 10. Higher figure indicates more pain. 10 is maximum pain.

CONTACTS AND LOCATIONS:
Overall Officials: Olof Wolf, Associate Professor, MD, Principal Investigator — Uppsala University Hospital and Uppsala University
Locations (11):
- Odense University Hospital, Odense, Denmark
- Tampere University Hospital, Tampere, Finland
- Østfold Hospital Trust, Fredrikstad, Norway
- Sweden (8):
  - Kalmar Regional Hospital, Kalmar
  - Linköping University Hospital, Linköping
  - Skane University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Danderyd Hospital, Stockholm
  - Stockholm South Hospital, Stockholm
  - Norrlands University Hospital, Umeå
  - Uppsala University Hopsital, Uppsala

IPD SHARING:
Plan to Share IPD: No